CLINICAL TRIAL: NCT01838057
Title: Evaluation of the Clinical and Economic Impact of Pfizer's painPRIMER Program in the Treatment of Low Back Pain in a Primary Care Setting
Brief Title: Evaluation of the Clinical and Economic Impact of painPRIMER in the Treatment of Low Back Pain in a Primary Care Setting
Status: Terminated | Type: Observational
Why Stopped: The study was terminated on 02-Jun-2014 due to slow enrollment. The study was not terminated for reasons of either safety or efficacy.
Sponsor: Pfizer (Industry)
Collaborators: Piedmont Healthcare System (Unknown)
Responsible Party: Sponsor
Other Study IDs: X9001010
Record Dates: First submitted 2013-04-15; First posted 2013-04-23 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- painPREMIER cohort
  Interventions: Device: painPREMIER cohort
- Control cohort
  Interventions: Other: Control cohort

INTERVENTIONS:
Device: painPREMIER cohort — Low back pain patients prospectively recruited during the study period and managed with painPREMIER.
  Groups: painPREMIER cohort
Other: Control cohort — A matched group of low back pain patients not managed with painPREMIER.
  Groups: Control cohort

SUMMARY:
To evaluate the impact of painPRIMER in a prospective six-month clinical investigation looking at clinical outcomes, health care professional and patient satisfaction, healthcare resource use, productivity and direct and indirect costs. The hypothesis is that early identification of the presence of neuropathic pain and back pain related comorbidities, to direct appropriate pharmacologic and non-pharmacologic treatment, painPRIMER would improve patient outcomes and reduce patient cycling, inappropriate use of imaging and surgery, thereby reducing costs and productivity loss associated with these inefficiencies.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 18 years of age
* Presenting to a HCP with low back pain
* Able to speak, write, and understand both verbal and written English

Exclusion Criteria:

* Conditions that may impede the patient's ability to participate in painPRIMER and complete the questionnaires, as per the HCP's discretion
* Patients presenting who have undergone surgery for back pain in the previous 12 months

  * Patients with Medicare as their primary insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with low back pain
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire: Change from baseline to month 3 in the Roland Morris Disability Questionnaire (RMDQ) total score in the painPRIMER cohort vs control cohort | 3 month
Low back pain (LBP) Cost: LBP (specific and related) direct medical costs associated with utilization of healthcare incurred by each study patient from baseline to month 6 | 6 month

SECONDARY OUTCOMES:
Change from baseline to month 6 in RMDQ total score | 3 and 6 months
Change from baseline to month 3 and 6 in low back pain intensity (LBPI) | 3 and 6 months
Change from baseline to month 3 and 6 daily sleep interference rating scale (DSIRS) | 3 and 6 months
Response as defined as a the proportion of patients with at least 30% and 50% improvement in LBPI at 3 and 6 months | 3 and 6 months
Response as defined as a the proportion of patients with at least 30% and 50% improvement in RMDQ at 3 and 6 months | 3 and 6 months
Quality of Life in the painPRIMER cohort vs control cohort: Change from baseline to month 3 and 6 in the Short- Form. | 3 and 6 months
psychosocial outcomes in the painPRIMER cohort and control cohort: Proportion of patients at risk for depression and/or anxiety (via Patient Health Questionnaire-4 [PHQ-4]) at baseline, 3 and 6 months | 3 and 6 months
psychosocial outcomes in the painPRIMER cohort and control cohort: Changes from baseline to month 3 and 6 in patients at risk for depression (PHQ-8) and anxiety (GAD-7), among those receiving the instrument (NOTE: only given to those scoring >/= | 3 and 6 months
3 on PHQ-4) | 3 and 6 months
psychosocial outcomes in the painPRIMER cohort and control cohort: Change from baseline to month 3 and 6 in catastrophizing (Coping Strategies Questionnaire -Catastrophizing [CSQ-CAT]) | 3 and 6 months
productivity/indirect costs: Changes from baseline to month 3 and 6 in Work Productivity and Activity Impairment (WPAI): Specific Health Problem, LBP | 3 and 6 months
Direct cost: Comparison of resource use/direct medical costs, in 6 months pre-enrollment/index date and 6 months post-enrollment/index date via insurance claims data for painPRIMER and control cohorts | 3 and 6 months
Patient satisfaction with painPRIMER | 3 and 6 months
Healthcare professional satisfaction with painPRIMER | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Fayetteville, Georgia, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=X9001010&StudyName=Evaluation%20of%20the%20Clinical%20and%20Economic%20Impact%20of%20%20painPRIMER%20in%20the%20Treatment%20of%20Low%20Back%20Pain%20in%20a%20Primary%20Care%20Setting%20